CLINICAL TRIAL: NCT07192497
Title: Therapeutic Effectiveness of Dry Needling and Acupressure Therapy Among Patients With Cervicogenic Headache
Acronym: headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Care Center (NHC) The Doctors Plaza Physical Therapy (Other)
Responsible Party: Principal Investigator, Atif Hussain, Principal investigator, Lincoln University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LUC/CPGS/PDFRA/PDA20250530/001; LUC/CPGS/PDFRA/PDA20250530/001 (Registry Identifier: PhD, health Sciences, Lincoln university college Malaysia)
Record Dates: First submitted 2025-07-18; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-06

CONDITIONS: Cervicogenic Headache
Keywords: cervical pain; Headache; Dry needling; Accupressure; myofascial trigger points
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain; Headache | interventions — Dry Needling; Acupressure

STUDY DESIGN:
Who Masked: Participant
Masking Description: only participants were unaware of treatment selection and choice of techniques would be applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A - Dry Needling (n=20) (Experimental): Dry needling at Myofascial trigger points
  Interventions: Other: DRY NEEDLING
- Group B- Acupressure (n=20) (Experimental): Manual pressure applied at cervical and shoulder acupressure points
  Interventions: Other: Acupressure
- Group C - Dry needling and Acupressure (n=20) (Experimental): Dry needling and acupressure therapy will be applied in the same session
  Interventions: Other: Dry needling and Acupressure therapy
- Control Group D - Hot Pack (n=20) (Experimental): Passive heat therapy applied to the cervical spine
  Interventions: Other: Hot Pack

INTERVENTIONS:
Other: DRY NEEDLING — Myofacial trigger point dry needling used to treat taught bands superficial or deep inside of muscles .
  Arms: Group A - Dry Needling (n=20)
Other: Acupressure — Acupressure therapy based on traditional Chinese principles
  Arms: Group B- Acupressure (n=20)
Other: Dry needling and Acupressure therapy — combination of dry needling and acupressure therapy on cervical trigger points
  Arms: Group C - Dry needling and Acupressure (n=20)
Other: Hot Pack — Hot fermentation will be applied on cervical pain area
  Arms: Control Group D - Hot Pack (n=20)

SUMMARY:
A randomized controlled trial (RCT) with a pre-test and post-test design will be conducted to compare the therapeutic effectiveness of Dry Needling (DN), Acupressure Therapy (AT), and their combination (DN + AT) against a control group receiving Hot Pack Therapy in patients diagnosed with Cervicogenic Headache (CH).

This study follows the CONSORT (Consolidated Standards of Reporting Trials) guidelines to ensure methodological transparency and rigor. The trial design includes:

* Randomization: Participants will be randomly assigned into four study groups.
* Blinding: A single-blind approach will be used, where participants are unaware of their group allocation, while the researchers administering the intervention will be aware.
* Follow-up Period: Pre-assessment at baseline, post-intervention assessment, and 2-week follow-up.
* Data Analysis: Standardized assessment tools will be used to evaluate the effectiveness of each intervention.

DETAILED DESCRIPTION:
Study Duration Total Duration: 1 year Intervention Period: 2 weeks Follow-Up: Pre-test, post-test, and 2-week follow-up Intervention Procedures

1. Group A (Dry Needling Therapy - DN)

   * 06 sessions over 2 weeks
   * Needling sites: Myofascial trigger points in cervical muscles
   * Session duration: 20-30 minutes
   * Post-treatment: Cryotherapy (5 minutes)
2. Group B (Acupressure Therapy - AT)

   * 06 sessions over 2 weeks
   * Pressure applied to cervical acupressure points
   * Post-treatment: Cryotherapy (10 minutes)
3. Group C (Combined Therapy - DN + AT)

   * 06 sessions over 2 weeks
   * Both DN and AT applied in sequence
   * Post-treatment: Cryotherapy (10-15 minutes)
4. Group D (Control - Hot Pack Therapy)

   * 06 sessions over 2 weeks
   * 15-minute heat therapy per session
   * No active intervention

ELIGIBILITY:
Inclusion Criteria:

Male and female patients aged 20 to 50 years Diagnosed with Cervicogenic Headache (CGH) based on International Headache Society (IHS) diagnostic criteria Chronic CGH symptoms (i.e., persisting for at least 3 months) No previous dry needling (DN) or acupressure therapy (AT) within the last 6 months Able and willing to provide informed consent and comply with treatment and follow-up protocols

Exclusion Criteria: History of cervical spine surgery, significant trauma, or vertebral tumors/neoplasms Congenital spinal deformities (e.g., scoliosis, spina bifida) Diagnosed with cervical radiculopathy, vestibular disorders, vertebrobasilar insufficiency, or cervical fractures Current use of anti-inflammatory drugs, muscle relaxants, or analgesics that may affect pain perception Diagnosed neurological, musculoskeletal, or orthopaedic conditions that affect balance, gait, or functional mobility Pregnancy (optional, often excluded in physiotherapy/dry needling trials)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Pain intensity (Numeric Pain Rating Scale, NPRS) | 04 weeks
  Pain intensity (Numeric Pain Rating Scale, NPRS) that is comprises over no's from 0 to 10 .
  0 consider as no pain while 10 considered as worst pain.

SECONDARY OUTCOMES:
secondary out come measures | A pre-test/post-test design with assessments at baseline and after two weeks of intervention. after 02 weeks intervention Week 3, and Week 4 for follow up total 02 weeks intervention and 02 weeks for followup
  Cervical range of motion
functional status | A pre-test/post-test design with assessments at baseline and after two weeks of intervention. after 02 weeks intervention Week 3, and Week 4 for follow up total 02 weeks intervention and 02 weeks for followup
  functional status by (Patient-Specific Functional Scale, PSFS).
Quality of life of patients with cervicogenic headache | A pre-test/post-test design with assessments at baseline and after two weeks of intervention. after 02 weeks intervention Week 3, and Week 4 for follow up total 02 weeks intervention and 02 weeks for followup
  impact on human Quality of life of patients with cervicogenic headache will be measured by using Headache Impact Test
Psycho-social characteristics | A pre-test/post-test design with assessments at baseline and after two weeks of intervention. after 02 weeks intervention Week 3, and Week 4 for follow up total 02 weeks intervention and 02 weeks for followup
  Psycho-social characteristics by (Depression, Anxiety, and Stress Scale-21, DASS-21
Sleep quality | A pre-test/post-test design with assessments at baseline and after two weeks of intervention. after 02 weeks intervention Week 3, and Week 4 for follow up total 02 weeks intervention and 02 weeks for followup
  Sleep quality by Pittsburgh Sleep Quality Index (PSQI

CONTACTS AND LOCATIONS:
Overall Officials: professor Dr. Sateesh babu Natarajan Supervisor, PhD, Study Director — Lincoln University College Malaysia
Locations (1):
- NHC(Doctors plaza physical therapy and Rehabilitation Centre), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to ethical considerations and the need to protect participant confidentiality, individual participant data will not be shared. The informed consent obtained from participants does not include permission for data sharing with external researchers.

REFERENCES:
- [Background] https://www.ncbi.nlm.nih.gov/books/NBK507862/
- See also: cervicogenic headache — https://www.nhc.net.pk/index.html